CLINICAL TRIAL: NCT06114849
Title: Analysis of a Peer-to-Peer Support Social Media Platform for Service Members and Veterans of the U.S. Military: Intervention 1 (Professional Outreach)
Brief Title: Brief Interventions on Social Media to Reduce Suicide Risk (Intervention 3)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment and enrollment. Unable to meet target N.
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Matthew Nock, Professor, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB19-1260-3
Record Dates: First submitted 2023-10-30; First posted 2023-11-02 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Suicide; Distress, Emotional
MeSH Terms: conditions — Suicide | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Participants will be identified using a machine learning risk algorithm developed by the investigators that will automatically identify concerning posts (e.g., those mentioning suicidal thoughts or behaviors). RallyPoint members whose posts are flagged will randomly be assigned to the intervention group or the control group.
  Interventions: Behavioral: Treatment as usual
- Intervention (Experimental): Participants will be identified using a machine learning risk algorithm developed by the investigators that will automatically identify concerning posts (e.g., those mentioning suicidal thoughts or behaviors). RallyPoint members whose posts are flagged will randomly be assigned to the intervention group or the control group.
  Interventions: Behavioral: Treatment as usual; Behavioral: Barrier Reduction Intervention

INTERVENTIONS:
Behavioral: Treatment as usual — Treatment-as-usual will follow the existing RallyPoint procedures for concerning posts on the site. In the current procedures, a RallyPoint staff member sends a supportive message to the member containing resource information on the Veteran's Crisis line, 911, and connecting with a therapist. This information is typically sent within 24 hrs of seeing a concerning post. Participants in both the control and intervention conditions will receive treatment-as-usual.
Behavioral: Barrier Reduction Intervention — After a post is identified in real-time by the risk algorithm, participants will be shown a pop-up message offering information on mental health resources (e.g., crisis line). Participants will be asked about their likelihood of using these resources. For participants who indicate they are not likely to use these resources, they will then be presented with a list of common barriers to help-seeking, drawing from research in this area (e.g., "Treatment is too expensive" or "I'm concerned about the police or paramedics getting involved."). Participants will be asked to click on any reason that resonates with them. When they click on a particular reason, they will then be presented with psychoeducational information to allay their concerns and encourage professional help-seeking.
  Arms: Intervention

SUMMARY:
This clinical trial is part of a series of brief interventions to reduce suicide risk in collaboration with the social media platform RallyPoint, a site specifically designed for U.S. servicemembers and veterans to connect with one another. In this RCT (Intervention 3: Professional Outreach), the investigators will test a psychoeducational intervention aimed at increasing users' likelihood of reaching out to mental health resources (e.g., suicide hotline) when experiencing distress.

DETAILED DESCRIPTION:
Both active duty and veterans of the United States military are at elevated risk for the development of psychological disorders such as depression, posttraumatic stress disorder, alcohol and substance use disorders, and suicide. Despite the clear need for psychological interventions for this population, only a small proportion of veterans utilize the Veteran's Affairs Health Care System for psychiatric care. Further, most people who are at-risk for suicide do not present for mental health treatment prior to their deaths. There are several reasons why military personnel may not seek out treatment, including stigma of mental health care, or structural barriers such as availability of treatment. Prior research from the current team comparing Army soldiers who died by suicide to matched control soldiers found that suicide decedents were more likely to perceive concerns that receiving mental health care would hurt their careers, reduce others' confidence in them, or lead others to see them as weak.

To increase the likelihood that veterans and servicemembers receive the help they need, one option is to harness technology to assess and treat mental health concerns outside of traditional healthcare settings. Social media platforms may be a particularly promising avenue for identifying and providing outreach to at-risk individuals, given research suggesting that peer support may be preferable to professional mental health treatment. In fact, a recent survey of military servicemembers conducted by the Defense Equal Opportunity Management Institute, servicemembers indicated that when they are feeling stressed, they prefer to speak with peers or spouses/partners (48-54%) rather than medical or mental health professionals (4-7%). Social media platforms may offer a scalable way of identifying and helping at-risk individuals.

In the current project, the investigators have partnered with the military-specific social media site RallyPoint (www.rallypoint.com) in order to determine how to best support at-risk veterans and servicemembers. The investigators will be testing three brief interventions aimed at connecting RallyPoint users to peer and professional resources:

Intervention 1: Peer support: This intervention will aim to improve RallyPoint users' ability to support their peers.

Intervention 2: Stigma-reduction intervention: This intervention will focus on reducing barriers that are inhibiting members in distress from reaching out to their peers.

Intervention 3: Professional Outreach (current intervention): This last intervention will aim to reduce barriers that are inhibiting members in distress from seeking professional mental health support.

ELIGIBILITY:
Inclusion Criteria:

* Active RallyPoint users who had at least one post flagged by a machine learning risk algorithm for containing concerning language (e.g., descriptions of suicidal thoughts or behaviors).

Exclusion Criteria:

* Active RallyPoint users who have not had any posts flagged by a machine learning risk algorithm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting use of resources | 24 hrs post intervention
  The investigators are primarily interested in whether participants in both groups contacted professional/emergency services after receiving the intervention or treatment-as-usual. Participants will be sent follow-up surveys to ask about which resources they have contacted.

CONTACTS AND LOCATIONS:
Locations (1):
- RallyPoint Networks, Inc, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No